CLINICAL TRIAL: NCT00667134
Title: Stimulatory Autoantibodies to the PDGFR and Phosphorylation of the PDGFR in Patients With Systemic Sclerosis
Brief Title: Stimulatory Autoantibodies to the Platelet-Derived Growth Factor Receptor (PDGFR) in Patients With Systemic Sclerosis
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Kristine Phillips, clinical assistant professor, University of Michigan
Other Study IDs: HUM00009559
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis autoantibodies
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — skin serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Subjects with diffuse scleroderma
- 2: Subjects with limited scleroderma
- 3: Subjects without a fibrosing or autoimmune disease.

SUMMARY:
This study is to determine if subjects with .systemic sclerosis have stimulatory autoantibodies to the PDGF receptor and to confirm activation (phosphorylation) of the PDGF receptor in skin sites with varying degrees of skin thickening

DETAILED DESCRIPTION:
Pilot study to assess whether patients with systemic sclerosis have stimulatory autoantibodies to the PDGF receptor and to confirm activation (phosphorylation) of the PDGF receptor in skin sites with varying degrees of skin thickening

ELIGIBILITY:
Inclusion Criteria:

1. Fulfill the American College of Rheumatology criteria for systemic sclerosis or:
2. Have no diseases that result in primary fibrosis of an organ system, including the skin and do not have an autoimmune disease

Exclusion Criteria:

1. If the subject has systemic sclerosis resulting from an environmental exposure
2. If the subject has an autoimmune disease excluding scleroderma
3. If the subject has an active infection (including, but not limited to hepatitis B, hepatitis C and HIV)
4. If the subject has been treated with cyclophosphamide in the past 8 weeks.
5. If the subject is prone to bleeding because they are on medications that thin the blood or have a low platelet count.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects from a tertiary care clinic specializing in scleroderma. Controls recruited by subjects being biopsied.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Stimulatory autoantibodies to the PDGF receptor | 1 year

SECONDARY OUTCOMES:
Phosphorylation of the PDGF receptor in patients with systemic sclerosis | One year

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Phillips, MD, Principal Investigator — University of Michigan; Julie A Konkle, BSN, Study Director — University of Michigan
Locations (1):
- University of Michigan Medical School, Ann Arbor, Michigan, United States